CLINICAL TRIAL: NCT02220283
Title: Comparison of the Effects of Open and Endovascular Aortic Aneurysm Repair on Long-term Renal Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201405032RINB
Record Dates: First submitted 2014-08-18; First posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Long-term Renal Dysfunction
Keywords: Acute kidney injury,aortic dissection
MeSH Terms: conditions — Acute Kidney Injury; Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Compare the renal complication of endovascular and open repair of acute aortic dissection by including patient treated at NTUH in 2010~2013.

ELIGIBILITY:
Patient underwent endovascular and open repair of aortic aneurysm at NTUH in 2010~2013 Age > 20 years old

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient underwent endovascular and open repair of aortic aneurysm at NTUH in 2010~2013
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Long-term change of renal function (eGFR) after operation of aortic aneurysm | 30 days

SECONDARY OUTCOMES:
Survival after operation of aortic aneurysm | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Fu Lai, MD, Principal Investigator
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan